CLINICAL TRIAL: NCT04587492
Title: Metabolome of Children With Spinal Muscular Atrophy Treated With Nusinersen
Brief Title: Metabolomics of Children With SMA
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Damjan Osredkar, Associate Professor in Pediatrics, University Medical Centre Ljubljana
Other Study IDs: 0120-305/2018/11
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy, nusinersen, metabolome
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid, serum, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with SMA: All children with SMA are eligible for the study
  Interventions: Drug: Nusinersen

INTERVENTIONS:
Drug: Nusinersen — Treatment with nusinersen

SUMMARY:
The aim of the proposed project is to evaluate whether the metabolome of patients with spinal muscular atrophy (SMA) before the initiation of treatment with nusinersen differs from the metabolome of healthy individuals and whether it changes 14 months after treatment with nusinersen.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a severe, debilitating disease and is an important source of morbidity and mortality of children. Novel disease modifying therapies can alter the natural course of the disease. However, many aspects of their action remain unknown. Metabolomics is the large-scale study of metabolites, within cells, biofluids, tissues or organisms. Collectively, these small molecules and their interactions within a biological system are known as the metabolome.

The aim of this study is to evaluate whether the metabolome of patients with SMA before the initiation of disease modifying therapy with nusinersen differs from the metabolome of healthy individuals. Next, we would like to asses whether tretament with nusinersen alters the metabolome of patients with SMA. Utilizing metabolomics, we would like to assess whether we can identify parameters reflecting the state of the disease in a particular patient, and parameters with diagnostic and/or prognostic value. Using metabolomics, we will aim to identify SMA patients that will positively respond to gene therapy.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed SMA
* Age up to 21 years

Exclusion Criteria:

* None

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with genetically diagnosed SMA
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Metabolomic difference from healthy children | Beginning of study
  Metabolomic difference between children with SMA and healthy children
Metabolomic change before and after treatment | At least 14 months of treatment
  Metabolomic change in children with SMA before and after treatment with nusinersen

CONTACTS AND LOCATIONS:
Locations (2):
- Slovenia (2):
  - Biotechnical faculty, Ljubljana
  - University Medical Centre Ljubljana, Ljubljana

IPD SHARING:
Plan to Share IPD: No